CLINICAL TRIAL: NCT00000676
Title: Randomized Comparative Study of Fluconazole Versus Clotrimazole Troches in the Prevention of Serious Fungal Infection in Patients With AIDS or Advanced AIDS-Related Complex. (A Nested Study of ACTG 081)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Purpose: Prevention
Other Study IDs: ACTG 981; 11504 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Candidiasis; Mycoses; HIV Infections
Keywords: Mycoses; Fluconazole; Clotrimazole; Antifungal Agents; Acquired Immunodeficiency Syndrome; AIDS-Related Complex
MeSH Terms: conditions — Candidiasis; Mycoses; HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Clotrimazole; Fluconazole

INTERVENTIONS:
Drug: Clotrimazole
Drug: Fluconazole

SUMMARY:
To study the effectiveness, safety, and tolerance of fluconazole versus clotrimazole troches (lozenges) as prophylaxis (preventive treatment) against fungal infections in patients enrolled in ACTG 081 (a study of prophylaxis against pneumocystosis, toxoplasmosis, and serious bacterial infection). Primarily, to compare the rates of invasive infections by C. neoformans, endemic mycoses, and Candida. To compare the mortality rates due to fungal infections between two antifungal prophylactic treatments. Secondarily, to assess the effect of prophylaxis on the incidence of severe fungal infections, defined as invasive infections and esophageal candidiasis and less severe mucocutaneous infection.

Serious fungal infections are significant complicating and life-threatening occurrences in patients with advanced HIV infection. Oropharyngeal candidiasis is found in almost all such patients, and causes pain, difficulty in swallowing, and loss of appetite. Similarly, esophageal candidiasis causes illness in the population. Cryptococcosis, endemic mycoses, and coccidioidomycosis also cause significant illness and death in AIDS patients. Once established, fungal infections in AIDS patients generally require continuous suppressive therapy because attempts at curing these infections are usually unsuccessful. Fluconazole has a number of characteristics that would make it a logical candidate to examine as a prophylactic agent in patients with advanced HIV infection. Animal studies have shown it to be prophylactic in models of candidiasis, cryptococcosis, histoplasmosis, and coccidioidomycosis. Initial experience in patients with active cryptococcal meningitis appears favorable, and studies of oropharyngeal candidiasis show it to be effective.

DETAILED DESCRIPTION:
Serious fungal infections are significant complicating and life-threatening occurrences in patients with advanced HIV infection. Oropharyngeal candidiasis is found in almost all such patients, and causes pain, difficulty in swallowing, and loss of appetite. Similarly, esophageal candidiasis causes illness in the population. Cryptococcosis, endemic mycoses, and coccidioidomycosis also cause significant illness and death in AIDS patients. Once established, fungal infections in AIDS patients generally require continuous suppressive therapy because attempts at curing these infections are usually unsuccessful. Fluconazole has a number of characteristics that would make it a logical candidate to examine as a prophylactic agent in patients with advanced HIV infection. Animal studies have shown it to be prophylactic in models of candidiasis, cryptococcosis, histoplasmosis, and coccidioidomycosis. Initial experience in patients with active cryptococcal meningitis appears favorable, and studies of oropharyngeal candidiasis show it to be effective.

AMENDED: 11/01/90 Sufficient numbers of patients will be enrolled from all centers starting at week 8 of participation in the parent study to achieve a total of 240 evaluable patients who will remain in the nested study for a maximum duration of 45 months. Enrollment will continue until all eligible and interested 081 patients are enrolled. Fungal prophylaxis will begin at the time of enrollment into the nested study and will continue until an efficacy or safety end point is reached, until withdrawal from the nested study, or until death.

Original design: Patients included are those already enrolled in ACTG 081. Patients are enrolled from all centers at either week 8, 12, 16, 20, 24, 28, or 32 of participation in the parent study. They are randomized to receive either oral fluconazole or clotrimazole troches. Prophylaxis continues until a serious fungal infection develops, the end of the parent study is reached (which is expected to be December 1991), the patient withdraws from either the nested or parent study, or the patient dies. Clinical examination is performed at 2 weeks and then monthly (or more if clinically indicated) for the duration of antifungal prophylaxis; the schedule of evaluation is the same as for the parent study. There is a 1-month postprophylaxis follow-up after discontinuation of prophylaxis for any reason.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* Zidovudine (AZT).
* Antipneumocystis prophylaxis.

Allowed:

* Topical suppressive antifungal agents.

Eligibility requirements are:

* Participation in NIAID ACTG 081.
* No history of systemic fungal infection, including esophageal or systemic candidiasis, cryptococcosis, histoplasmosis, coccidioidomycosis, blastomycosis, sporotrichosis, or aspergillosis.
* Willingness to sign an informed consent.
* Transaminases < 5 x upper limit of normal.
* Noncompliance will not be a reason for withdrawal of a patient from the study, unless patient refuses further treatment.

Allowed:

* A history of oropharyngeal, vaginal or cutaneous candidiasis.
* Dermatophyte infections (i.e., tinea pedis) at entry but not active candida infection. Sites of suspected dermatophyte involvement other than the feet should have candida excluded by culture.

Prior Medication:

Allowed:

* Topical suppressive antifungal agents.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or diseases are excluded:

* History of systemic fungal infection, including esophageal or systemic candidiasis, cryptococcosis, histoplasmosis, coccidioidomycosis, blastomycosis, sporotrichosis, or aspergillosis.
* Active systemic fungal infection at time of enrollment.
* Active superficial fungal infection at time of entry. (Such patients may be treated with topical antifungal agents and may be randomized if they are in clinical remission 14 days after completion of such therapy.)

Concurrent Medication:

Excluded:

* Amphotericin B.
* Fluconazole.
* Itraconazole.
* SCH 39304.
* Other systemic antifungals.

Patients with the following are excluded:

* Previous or currently active systemic fungal infection.
* History of allergy or intolerance to imidazole or azoles.
* Positive serum cryptococcal antigen titer at any dilution.
* Requiring multi-agent therapy for tuberculosis or for symptomatic Mycobacterium avium infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Study Completion 1993-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bozzettee S, Study Chair; Powderly WG, Study Chair
Locations (26):
- United States (25):
  - Stanford CRS, Palo Alto, California
  - Ucsd, Avrc Crs, San Diego, California
  - Ucsf Aids Crs, San Francisco, California
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Northwestern University CRS, Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Tulane Med. Ctr. - Charity Hosp. of New Orleans, ACTU, New Orleans, Louisiana
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Bmc Actg Crs, Boston, Massachusetts
  - Beth Israel Deaconess - East Campus A0102 CRS, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - Washington U CRS, St Louis, Missouri
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - Memorial Sloan-Kettering Cancer Ctr., New York, New York
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - Pitt CRS, Pittsburgh, Pennsylvania
  - University of Washington AIDS CRS, Seattle, Washington
- Mbeya Med. Research Program, Mbeya Referral Hosp. CRS, Mbeya, Tanzania

REFERENCES:
- [Background] Glick ME. CTG studies yield results. AIDS Clinical Trials Group. NIAID AIDS Agenda. 1995 Spring:8-9. PMID 11362451
- [Background] Hanna L. Treatment for HIV-related fungal infections. BETA. 1995 Jun:10-7. PMID 11362539
- [Background] Powderly WG. Fungal infections. Program Abstr Intersci Conf Antimicrob Agents Chemother. 1994 Oct 4-7:274
- [Background] Powderly WG. Prophylaxis of fungal infection in HIV infection. Program Abstr Intersci Conf Antimicrob Agents Chemother. 1994 Oct 4-7:270
- [Background] Powderly WG, Finkelstein D, Feinberg J, Frame P, He W, van der Horst C, Koletar SL, Eyster ME, Carey J, Waskin H, et al. A randomized trial comparing fluconazole with clotrimazole troches for the prevention of fungal infections in patients with advanced human immunodeficiency virus infection. NIAID AIDS Clinical Trials Group. N Engl J Med. 1995 Mar 16;332(11):700-5. doi: 10.1056/NEJM199503163321102. PMID 7854376